CLINICAL TRIAL: NCT02385929
Title: Bimodal Pre-habilitation Program to Improve Symptom Control After Treatment for Head and Neck Cancer
Brief Title: Pre-habilitation of Patients With Head and Neck Cancer
Acronym: SYNK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Irene Wessel (Other)
Collaborators: Danish Cancer Society (Other); Danish Association of Occupational Therapist (Other); Rigshospitalet, Denmark (Other); Danish Cancer Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Irene Wessel, Consultant, ph.d., associate professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-2-2014-074; R108-A6969-14-S31 (Other Grant/Funding Number: The Danish Cancer Society)
Record Dates: First submitted 2015-02-09; First posted 2015-03-11 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Intervention; Rehabilitation; Late Effects; Dysphagia
MeSH Terms: conditions — Head and Neck Neoplasms; Deglutition Disorders | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swallowing therapy & resistance training (Experimental): Mouth opening and swallowing exercise intervention by occupational therapist for half an hour 3 times a week for 5-6 weeks during radiotherapy.
  Progressive resistance training by physiotherapist for 1 hour twice weekly for 5-6 weeks during radiotherapy.
  Interventions: Behavioral: Swallowing therapy & resistance training
- Standard Care (No Intervention): Patients in this arm are randomized to usual care / control group

INTERVENTIONS:
Behavioral: Swallowing therapy & resistance training — i) Individual instructions in swallowing and mouth opening exercises 3 days per week by occupational therapist throughout radiotherapy, ii) Progressive resistance training twice weekly by physiotherapist, either individually or group based, throughout radiotherapy, iii) Daily home-based swallowing and mouth opening exercises from beginning of treatment until 2 months after end-of-treatment.
  iv) Weekly follow-up phone contacts with occupational therapists from end-of-treatment and 2 months onwards.
  Arms: Swallowing therapy & resistance training

SUMMARY:
The purpose of this study is to explore whether early initiated physical exercise concurrent with a swallowing and mouth opening exercise program will have a positive effect on swallowing function and other quality of life aspects in patients treated with radiotherapy for head and neck cancer. The investigators hypothesize that patients who complete the program will have improved swallowing function and physical function one year after completing their treatment compared to patients who do not participate in the training program.

DETAILED DESCRIPTION:
Although the potential negative impact of head and neck cancer (HNC) and its treatment on eating ability and quality of life is well documented there is no evidence based and standardized rehabilitation program available for Danish patients affected by HNC while going through radiotherapy (with or without concurrent chemotherapy). This study proposal is based on a thorough literature review on HNC treatment and late effects, and interventions targeting dysphagia and physical functioning.

Traditionally, rehabilitation is initiated when loss of function is already established. Emerging evidence suggests, however, that it can be of benefit to the patient to initiate an early rehabilitation process (prehabilitation) starting before initiation of treatment and during treatment. Prehabilitation aims to enhance pre-treatment functional capacity for better tolerance of treatment, facilitate general recovery, and prevent development of functional impairment or reduce the extent of these problems in a long-term perspective. HNC patients have a unique set of functional challenges such as pre- and post-treatment dysphagia, pain, and weight loss and often also high baseline levels of alcohol and tobacco consumption. In addition, studies have shown that only 31 % and 9 % of HNC patients are meeting public health guidelines for physical activity before and after diagnosis, respectively, and that weight loss in HNC patients treated with chemoradiation begin after only 1 week of therapy. Most of the weight loss was lean body mass (LBM) rather than fat loss. Loss of LBM is significantly associated with physical performance and increased functional dependence. The level of physical activity typically decreases significantly during treatment.

Dysphagia is considered the most prominent complication to HNC and its treatment, affecting physical function and quality of life. Post treatment dysphagia occurs in a significant proportion of patients and results from multiple factors such as xerostomia, taste loss, decreased sensory function, fibrosis and trismus. Disuse of swallowing muscles due to acute radiation effects or tube feeding can contribute to decline in swallowing function. Often, difficulties in swallowing and mouth opening are presenting features of HNC even at the time of diagnosis. To reduce these problems, patients may do a series of exercises before and during treatment to promote strength, mobility, and endurance of base of tongue, pharyngeal constrictors, and suprahyoid strap muscles. Although no definitive trials have yet been carried out, small randomized controlled trials (RCTs) and observational studies investigating pre-treatment swallowing and/or mouth opening exercise programs show promising benefits. Further, the few studies of resistance and cardio training on functional capacity in HNC patients are generally promising with medium to large effects on fatigue and physical function measures. For weight loss it seems as if progressive resistance training (PRT) is able to almost reverse the loss of LBM in HNC patients.

Generally studies on swallowing therapy for HNC patients have relied greatly on self-practice, and thus report low compliance. In view of this knowledge the investigators determine that there is a need for studies that include patients with HNC undergoing (chemo)radiation therapy focusing on i) prevention of dysphagia and loss of muscle strength and ii) improvement of compliance to mouth opening and swallowing exercises.

The purpose of the SYNK study is a randomized design to test the effect of theory based intervention on eating dysfunctions secondary to radiation treatment for HNC. The SYNK intervention consists of: i) individual instructions in swallowing and mouth opening exercises 3 days per week by occupational therapist throughout radiotherapy, ii) progressive resistance training twice weekly by physiotherapist, either individually or group based, throughout radiotherapy, iii) daily home-based swallowing and mouth opening exercises from beginning of treatment until 2 months after end-of-treatment (self-practice), and iv) weekly follow-up phone contacts with occupational therapists from end-of-treatment and 2 months onwards.

The investigators will enroll patients from the Oncological Department Rigshospitalet and randomize 240 patients. Patients will be randomized (1:1) to standard care plus the SYNK intervention and to standard care (control group).

The proposed study has the potential to support the general health status of HNC patients as well as to minimize adverse late effects of treatment (i.e. swallowing and mouth opening difficulties, general physical deterioration due to physical inactivity and problems with eating, and reduced QoL). The design of the intervention, being early, intensive and bimodal adds a new dimension to research in the prevention of devastating late effects in this particularly vulnerable patient group.

The investigators hypothesize that the SYNK intervention will:

* Improve swallowing function
* Improve physical function to stop the loss of muscle strength
* Improve quality of life and lessen the symptoms of anxiety and depression

ELIGIBILITY:
Inclusion Criteria:

* Histological proven cancer in one or more of the following areas: larynx, hypopharynx, oropharynx, cavi oris, or unknown primary tumor
* Set to curative radiotherapy with or without concurrent chemotherapy for treatment of cancer in the head and neck region in accordance with the Danish Head and Neck Cancer Group (DAHANCA) guidelines
* Fully self-reliant
* Danish skills, oral and written
* Informed consent

Exclusion Criteria:

* Previously received treatment for head and neck cancer (radiotherapy, chemotherapy and/or surgery).
* Pregnancy
* ECOG performance status > 2
* Presence of psychological-, family-, sociological- or geographical issues that could prevent the patient from completing the intervention
* Simultaneous or previous illness or conditions that could prevent the patient's ability to complete the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Swallowing function measured by penetration aspiration scale (PAS) during a Fiber Endoscopic Evaluation of Swallowing (FEES). | Baseline, 14 weeks and 58 weeks. Participants will be followed up till 12 months after they finalize their radiotherapy, an expected average of 58 weeks from baseline.
  To investigate the change in swallowing function among patients in intervention- and the control group from baseline to 14 and 58 weeks follow up and the difference in change between intervention - and the control group.

SECONDARY OUTCOMES:
Level of fatigue by the EORCT QLQ-C30 3-point fatigue subscale. | baseline, 6 weeks, 14 weeks, 28 weeks and 58 weeks.
  To investigate the change in fatigue among patients in intervention- and the control group from baseline to 6,14, 28 and 58 weeks follow up and the difference in change between intervention - and the control group.
Maximal Interincisal Distance (MID) by Therabite Range of Motion (ROM) scale | baseline, 6 weeks, 14 weeks, 28 weeks and 58 weeks.
  To investigate the change in mouth opening and the development of trismus (defined as MID ≤ 35mm) among patients in intervention- and the control group from baseline to 6,14, 28 and 58 weeks follow up and the difference in change between intervention - and the control group.
Dysphagia related quality of life by M.D. Anderson Dysphagia Inventory (MDADI) | baseline, 6 weeks, 14 weeks, 28 weeks and 58 weeks.
  To investigate the change in patient reported quality of life related to dysphagia among patients in intervention- and the control group from baseline to 6, 14, 28 and 58 weeks follow up and the difference in change between intervention - and the control group. We will also use this outcome to evaluate correlation or deviations in patient vs observer rated outcomes by comparing the MDADI to the PAS score (primary outcome).
Health related quality of Life by the European Organisation for Research and Treatment of Cancer (EORCT) Quality if Life Questionnaire (QLQ)-30 and EORCT QLQ - H&N35 | baseline, 6 weeks, 14 weeks, 28 weeks and 58 weeks.
  To investigate the change in health related quality of life among patients in intervention- and the control group from baseline to 6,14, 28 and 58 weeks follow up and the difference in change between intervention - and the control group.
Level of oral intake by Functional Oral Intake Scale (FOIS) | baseline, 6 weeks, 14 weeks, 28 weeks and 58 weeks.
  To investigate the change in oral intake and tube dependency among patients in intervention- and the control group from baseline to 6,14, 28 and 58 weeks follow up and the difference in change between intervention - and the control group.
Weight loss by body weight | baseline, 6 weeks, 14 weeks, 28 weeks and 58 weeks.
  To investigate the change in weight loss among patients in intervention- and the control group from baseline to 6,14, 28 and 58 weeks follow up and the difference in change between intervention - and the control group.
Physical strength by 30 seconds Sit to Stand (STS) test. | baseline, 6 weeks, 14 weeks, 28 weeks and 58 weeks.
  To investigate the change in lower extremities' strength as an expression of the overall physical strength among patients in intervention- and the control group from baseline to 6,14, 28 and 58 weeks follow up and the difference in change between intervention - and the control group.
Pain by numerical rating scale (NRS) | baseline, 6 weeks, 14 weeks, 28 weeks and 58 weeks.
  To investigate the change in pain among patients in intervention- and the control group from baseline to 6,14, 28 and 58 weeks follow up and the difference in change between intervention - and the control group.
Depression by Major Depression Inventory (MDI) | baseline, 6 weeks, 14 weeks, 28 weeks and 58 weeks.
  To investigate the change in depressive symptoms among patients in intervention- and the control group from baseline to 6,14, 28 and 58 weeks follow up and the difference in change between intervention - and the control group.
Anxiety by Symptom Check List (SCL-92) Anxiety subscale | baseline, 6 weeks, 14 weeks, 28 weeks and 58 weeks.
  To investigate the change in anxiety among patients in intervention- and the control group from baseline to 6,14, 28 and 58 weeks follow up and the difference in change between intervention - and the control group.
Performance Status by Eastern Cooperative Oncology Group (ECOG) performance scale | baseline, 6 weeks, 14 weeks, 28 weeks and 58 weeks.
  To investigate the change in performance status among patients in intervention- and the control group from baseline to 6,14, 28 and 58 weeks follow up and the difference in change between intervention - and the control group.
Subjective symptoms of dysphagia by Eating Assessment Tool (EAT-10) | Participants will be followed up till 12 months after they finalize their radiotherapy, an expected average of 58 weeks from baseline.
  EAT-10 is a questionnaire screening tool used to evaluate patient-experienced symptoms of dysphagia and measures the level of ten specific difficulties related to swallowing. We will measure this outcome at the same time as our primary outcome to analyze the correlation between the subjective and objective measures of oropharyngeal dysphagia.

CONTACTS AND LOCATIONS:
Overall Officials: Sara F Hajdú, M.Sc, Principal Investigator — Rigshospitalet, Denmark; Susanne O Dalton, professor, Principal Investigator — Danish Cancer Society; Christoffer Johansen, professor, Principal Investigator — Rigshospitalet, Denmark; Irene Wessel, MD, phd, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Næstved Sygehus, Næstved, Region Sjælland
  - Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hajdu SF, Wessel I, Johansen C, Kristensen CA, Kadkhoda ZT, Plaschke CC, Dalton SO. Swallowing therapy and progressive resistance training in head and neck cancer patients undergoing radiotherapy treatment: randomized control trial protocol and preliminary data. Acta Oncol. 2017 Feb;56(2):354-359. doi: 10.1080/0284186X.2016.1269193. PMID 28206871
- [Background] Hajdu SF, Plaschke CC, Johansen C, Dalton SO, Wessel I. Cross-Cultural Translation, Adaptation and Reliability of the Danish M. D. Andeson Dysphagia Inventory (MDADI) in Patients with Head and Neck Cancer. Dysphagia. 2017 Aug;32(4):472-479. doi: 10.1007/s00455-017-9785-3. Epub 2017 Mar 7. PMID 28271296
- [Background] Fredslund SV, Hogdal N, Christensen MB, Wessel I. Dysphagia training after head and neck cancer fails to follow legislation and national recommendations. Dan Med J. 2015 May;62(5):A5067. PMID 26050828
- [Derived] Hajdu SF, Christensen MB, Kristensen MO, Wessel I, Johansen C, Dalton S. Adherence to preventive swallowing exercises for head and neck cancer patients undergoing (chemo)radiotherapy treatment. Acta Oncol. 2019 May;58(5):658-664. doi: 10.1080/0284186X.2018.1563715. Epub 2019 Jan 30. PMID 30698049